CLINICAL TRIAL: NCT04975165
Title: Comparison of Smart-phone Based Gait Analysis Between Simultaneous and Staged Total Knee Arthroplasties
Brief Title: Comparison of Gait Pattern Between Simultaneous and Staged Knee Arthroplasties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Deniz CANKAYA, Assoc. Professor, Gulhane Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/16
Record Dates: First submitted 2021-07-21; First posted 2021-07-23 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Bilateral Knee Osteoarthritis
Keywords: Bilateral knee arthroplasty; Gait analysis; Smart-phone
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staged total knee arthroplasty (Experimental): Staged replacement of both knees in two separate surgeries.
  Interventions: Procedure: Total knee arthroplasty
- Simultaneous total knee arthroplasty (Experimental): Simultaneous replacement of both knees in a single surgery.
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Bilateral surgery in one arm and staged surgery in another arm during total knee arthroplasty

SUMMARY:
Total knee arthroplasty is a well-known treatment of the end-stage osteoarthritis of the knee. In the case of bilateral end-stage knee osteoarthritis, both of the knees need total knee arthroplasty. Bilateral total knee arthroplasty could be performed simultaneously or staged according to the preference of the patients. Simultaneous total knee arthroplasty is defined as the replacement of both knees in a single surgery. The major advantage of simultaneous total knee arthroplasty this surgery is that it requires only one hospital stay and a rehabilitation period to recover both knees, but higher blood transfusion rates and thromboembolism risk are still major concerns. Therefore, in this comparative study, smart-phone based gait analysis and patient-reported functional outcomes are evaluated in patients undergoing simultaneous and staged total knee arthroplasty, at 3, 6, and 12 months postoperatively

DETAILED DESCRIPTION:
Patients with bilateral end-stage knee osteoarthritis will be included in the current study. Bilateral total knee arthroplasty will be performed simultaneously or staged according to the preference of the patients. We will have two groups: staged total knee arthroplasty and simultaneous total knee arthroplasty groups. The patients will be evaluated preoperatively and at 3, 6, and 12 months postoperatively, with knee scores (Knee Society Scores and Knee Injury and Osteoarthritis Outcome Score), life quality (SF-12), and smart-phone based gait analysis. All data will be calculated as mean and standard deviation values. The Student's t-test will be used for statistical analysis of the patient data. Statistical calculations will be performed using SPSS vn.22.0 software (IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of bilateral primary knee osteoarthritis Age 55 to 85 years Must be able to walk without support

Exclusion Criteria:

Rheumatological joint diseases Previous knee surgery Neuromuscular diseases Unilateral knee osteoarthritis Insufficiency of knee collateral ligaments.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
smart-phone based gait analysis | Change from preoperative gait analysis at 3rd month gait analysis
  Gait analysis (The gait velocity, step time (ST), step length (SL), cadence, step length symmetry and step time symmetry) is made using the Gait Analyzer version 0.9.95.0 (Control One LLC, NM, USA) smartphone application
smart-phone based gait analysis | Change from 3rd month gait analysis at 6th month gait analysis
  Gait analysis (The gait velocity, step time (ST), step length (SL), cadence, step length symmetry and step time symmetry) is made using the Gait Analyzer version 0.9.95.0 (Control One LLC, NM, USA) smartphone application
smart-phone based gait analysis | Change from 6th month gait analysis at 12th month gait analysis
  Gait analysis (The gait velocity, step time (ST), step length (SL), cadence, step length symmetry and step time symmetry) is made using the Gait Analyzer version 0.9.95.0 (Control One LLC, NM, USA) smartphone application

SECONDARY OUTCOMES:
Knee functional scores | Change from preoperative Knee Society Scores (KSS) at 3rd month Knee Society Score (KSS)
  Knee Society Score (KSS) (has two different subscale : Knee and Function 100-80: Excellent 79-70:Good 69-60:Fair below 60:Poor )
Knee functional scores | Change from 3rd month Knee Society Scores (KSS) at 6th month Knee Society Score (KSS)
  Knee Society Score (KSS) (has two different subscale : Knee and Function 100-80: Excellent 79-70:Good 69-60:Fair below 60:Poor )
Knee functional scores | Change from 6th month Knee Society Scores (KSS) at 12th month Knee Society Score (KSS)
  Knee Society Score (KSS) (has two different subscale : Knee and Function 100-80: Excellent 79-70:Good 69-60:Fair below 60:Poor )

CONTACTS AND LOCATIONS:
Overall Officials: Deniz CANKAYA, Assoc.Prof., Study Chair — Gulhane Teaching and Research Hospital
Locations (1):
- Gulhane Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No